CLINICAL TRIAL: NCT01899976
Title: A Non-Randomized, Multi-Center, Prospective, Single Arm Clinical Study of the X-SUIT NIR® Covered Biliary Metallic Stent for Palliation of Malignant Strictures in the Biliary Tree Via Endoscopic Approach
Brief Title: X-MAS Biliary Study With Covered Biliary Stent
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medinol Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Protocol Number BI-03-01
Record Dates: First submitted 2013-07-08; First posted 2013-07-16 (Estimated); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Biliary Tract Cancer
Keywords: covered biliary stent; X-Suit NIR Covered Biliary Stent; malignant strictures in biliary tree
MeSH Terms: conditions — Biliary Tract Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- X-Suit NIR Covered Biliary Stent (Other): Stent implantation in the biliary tree
  Interventions: Device: X-Suit NIR Covered Biliary Stent

INTERVENTIONS:
Device: X-Suit NIR Covered Biliary Stent

SUMMARY:
The purpose of this study is to provide safety and efficacy data for the X-Suit NIR® Covered Biliary Metallic Stent for subjects with malignant stricture(s) in the biliary tree. The study is designed to support the regulatory requirement of a 510(k) marketing application in the United States.

DETAILED DESCRIPTION:
This is a non-randomized, multi-center, prospective, single arm clinical study of the X-Suit NIR® Covered Biliary Metallic Stent for the palliation of malignant strictures in the biliary tree via endoscopic approach.

Adult males and females (≥ 18 years old), with clinical symptoms of biliary obstruction and inoperable extrahepatic biliary obstruction by any malignant process.

The expected duration of this study is approximately 18 months from the time of first subject enrollment to the time of the last subject's 6-month post stent implantation follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older.
2. Clinical symptoms of biliary obstruction.
3. Presence of inoperable extrahepatic distal biliary obstruction by any malignant process (the subject not being a surgical candidate based on the finding of a pancreatic mass >2.0cm or a severe medical illness).
4. Subject is willing and able to comply with the study procedures and provide written informed consent to participate in the study.
5. Insured by Social Security (applicable to subjects screened in France).

Exclusion Criteria:

* 1. Participation in an Investigational Study within 90 days prior to date of subject consent.

  2. Perforation of any duct within the biliary tree. 3. Presence of more than one previously implanted plastic stent. 4. Previous plastic stent implantation less than 2 weeks prior to current procedure.

  5. Presence of a metal biliary stent. 6. Presence of any esophageal or duodenal stent. 7. Previous Bilroth II or Roux-en-Y gastric resection, a significant duodenal obstruction or any other altered anatomy which could prevent access to ampulla.

  8. Subjects for whom endoscopic procedures are contraindicated. 9. Subjects with known sensitivity to any components of the stent or delivery system.

  10. Subjects with active hepatitis or other hepatic diseases that may cause jaundice.

  11. Subjects with a WHO performance score of 4 - Bedbound (completely disabled, cannot carry on any self-care, totally confined to bed or chair).

  12. Subjects known to be pregnant.

Cholangiographic exclusion criterion:

13. Strictures that cannot be passed by the guide wire or the delivery system.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2013-08; Primary Completion 2017-11-13 (Actual); Study Completion 2017-11-13 (Actual)

PRIMARY OUTCOMES:
Maintenance of a total serum bilirubin level ≤ 3.0 mg/dL or a reduction of >30% if baseline value was greater than 3.0 mg/dL | 6 months follow up or prior to death, whichever comes first
  Maintenance of a total serum bilirubin level ≤ 3.0 mg/dL or a reduction of >30% if baseline value was greater than 3.0 mg/dL- outcome

SECONDARY OUTCOMES:
total number of adverse events | 6 months
  total number of adverse events (anticipated and unanticipated)

CONTACTS AND LOCATIONS:
Overall Officials: Peter D Siersema, Prof., Principal Investigator — University Medical Center Utrecht, Netherlands
Locations (9):
- Hôpital Erasme Brussels (ULB), Brussels, Belgium
- Israel (6):
  - Hillel Yafeh Medical Center, Hadera
  - Rambam Medical Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Haddasah Medical Center, Jerusalem
  - Sheba Medical Center, Tel Hashomer, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Netherlands (2):
  - University Medical Center Utrecht, Utrecht, Heidelberglaan
  - Academic Medical Center (AMC), Amsterdam